CLINICAL TRIAL: NCT03228381
Title: An Acute Evaluation of Anatomical and Geometric Changes Using the Bladder on a Stick System (BOSS)
Brief Title: The BOSS Study: An Acute Evaluation of Anatomical and Geometric Changes Using the Bladder on a Stick System (BOSS)
Acronym: BOSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mardil Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: BOSS CT005
Record Dates: First submitted 2017-07-17; First posted 2017-07-24 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-04

CONDITIONS: Functional Mitral Regurgitation; Heart Failure
Keywords: Functional Mitral Regurgitation; Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- BOSS Device (Experimental): Patients who are undergoing open chest cardiac surgery via sternotomy will receive the BOSS device to assess acute anatomical and geometric annular and ventricular changes that occur when strategically positioned an external inflatable chambers are applied to the outside of the heart.
  Interventions: Device: BOSS Device

INTERVENTIONS:
Device: BOSS Device — The BOSS will be comprised of a flexible, medical grade silicone handle and interchangeable inflatable medical grade silicone chambers. The inflatable chambers will vary in geometry and will have silicone tubing attached to them to allow inflation and deflation of the chamber while in the pericardial space. During open chest cardiac surgery, a small incision will be made in the pericardium to allow for insertion of the BOSS device into the pericardial space. Once inserted, the BOSS device will be positioned in different locations around the outside of the heart and anatomical and geometric changes will be observed echocardiographically. Use of the BOSS device is expected to lengthen the procedure by an average of 15 minutes, and in rare instances may be extended beyond 15 minutes as deemed appropriate by the investigator. The BOSS will be removed prior to continuing with the planned surgery.

SUMMARY:
The objective of the BOSS Study is to assess acute anatomical and geometric annular and ventricular changes that occur when strategically positioned an external inflatable chambers are applied to the outside of the heart.

DETAILED DESCRIPTION:
Mardil Medical is developing an investigational device for functional mitral regurgitation intended to provide ventricular support with adjustable inflatable chambers to reduce annular dilation, correct papillary muscle displacement, and restore mitral valve leaflet coaptation. In doing so, Mardil Medical is interested in exploring the anatomical and geometric annular and ventricular changes that occur when strategically positioned external inflatable chambers are applied to the outside of the heart. Favorable benefits of circumferential reduction in ventricular wall stress favoring left ventricular (LV) remodeling and acute reshaping of LV segments subtending the deformed mitral valve apparatus needs to be better understood. Mardil Medical is pursuing this study as an initial phase in the Acute Evaluation of Anatomical and Geometric Changes using the Bladder on a Stick System (BOSS).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* Patient undergoing open chest cardiac surgery via sternotomy
* Signed informed consent by patient or legally authorized representative

Exclusion Criteria:

* Any procedure, condition or cardiac anatomy that may impact or compromise the pericardial space (e.g. prior valve surgery, CABG, epicardial pacing leads, pericarditis, history of mantle radiation, or other procedure involving pericardial access)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-08-21 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Acute anatomical changes assessed by echocardiography | At Procedure
  Anatomical annular and ventricular changes assessed by echocardiography, such as shape and deformation of the mitral valve annulus and left ventricular wall
Acute geometric changes measured by echocardiography | At Procedure
  Geometric annular and ventricular changes measured by echocardiography, such as reductions in septal-lateral dimension and left ventricular end diastolic diameter (LVEDD)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Hase, Study Director — Mardil Medical
Locations (3):
- United States (2):
  - Henry Ford Health System, Detroit, Michigan
  - Minneapolis Heart Institute at Abbott Northwestern Hospital, Minneapolis, Minnesota
- Sanatorio Italiano, Asunción, Paraguay

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers.